CLINICAL TRIAL: NCT06732466
Title: Clinical Research Study to Evaluate the Effect of a Toothpaste Containing Chlorhexidine 0.3% in Subjects With Established Dental Plaque and Gingivitis
Brief Title: Evaluation of the Effect of a Toothpaste Containing 0.3% Chlorhexidine in Subjects With Established Dental Plaque and Gingivitis
Acronym: CHX TP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2024-11-PG-CHX-BZ-CB
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: Gingivitis; Gingivitis and Periodontal Diseases; Gingival Disease; Dental Plaque
Keywords: chlorhexidine; toothpastes; gingivitis; dental plaque
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Gingival Diseases; Dental Plaque | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Phase III, one-center, parallel group, double blind and randomized trial
Who Masked: Participant, Investigator
Masking Description: In this clinical trial, masking involves several key roles to ensure unbiased results. The participant and the investigator are masked in this double-blind study. This means that the participants do not know which group they have been assigned to and the investigators conducting the study do not know the group assignments. This comprehensive masking approach is designed to minimize any potential biases and maintain the integrity of the study results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.3% chlorhexidine toothpaste (Experimental): Test group assigned to use a 0.3% chlorhexidine + 3% AmCl toothpaste and brushing with a commercially available adult soft bristle toothbrush
  Interventions: Drug: Chlorhexidine toothpaste; Device: Toothbrush
- Negative Control (Placebo Comparator): Negative Control group assigned to use a placebo toothpaste without chlorhexidine and AmCl and brushing with a commercially available adult soft bristle toothbrush
  Interventions: Device: Toothbrush; Drug: Placebo toothpaste without chlorhexidine and AmCl

INTERVENTIONS:
Drug: Chlorhexidine toothpaste — A toothpaste containing 0.3% chlorhexidine + 3% AmCl
  Arms: 0.3% chlorhexidine toothpaste
Device: Toothbrush — Commercially available adult soft bristle toothbrush
Drug: Placebo toothpaste without chlorhexidine and AmCl — Negative Control Group assigned to use a placebo toothpaste without chlorhexidine and AmCl and brushing with a commercially available adult soft bristle toothbrush.
  Arms: Negative Control

SUMMARY:
This is a Phase III, one-center, parallel group, double blind, clinical study to evaluate the effect of a toothpaste containing 0.3% chlorhexidine in subjects with established dental plaque and gingivitis. It involves 80 participants aged between 18 and 70, randomly assigned to different groups, and spans 21 days.

DETAILED DESCRIPTION:
This clinical study aims to evaluate the effect of a toothpaste containing 0.3% chlorhexidine in subjects with established dental plaque and gingivitis. It is a Phase III study designed as randomized, one-center, double blind, parallel group trial involving 80 participants aged 18 to 70. Subjects will be divided into two groups: test group - subjects assigned to use a toothpaste with a 0.3% chlorhexidine + 3% AmCl and brush with a commercially available adult soft bristle toothbrush; negative control group - subjects assigned to use a placebo toothpaste without chlorhexidine and AmCl and brush with a commercially available adult soft bristle toothbrush. Subjects will undergo baseline, 14 days and 21 days evaluations. The primary outcome will be reduction of gingival inflammation and data will be analyzed using ANCOVA to assess the efficacy of the test product. Adverse events and compliance will be closely monitored, with strict confidentiality maintained for all participants. The study rigorous design aims to provide comprehensive insights into the effectiveness of the chlorhexidine toothpaste regarding gingivitis and dental plaque control.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, between 18-70 years of age;
* Availability for the duration of the study;
* Good general health (absence of any condition that, in the opinion of the Principal Investigator, might constitute a risk to the subject while participating in the study. Examples include heart problems, valve/hip replacements, etc);
* Willingness to provide information related to their medical history;
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars and crowns);
* Initial gingivitis index a minimum average score of 1.5 as determined by the use of the Löe and Silness Gingival Index;
* More than 30% of bleeding sites and absence of periodontal disease;
* Informed Consent Form signed.

Exclusion Criteria:

* Absence of visible clinical signs of periodontal disease, such as the presence of suppuration, dental mobility, and/or extensive attachment loss;
* That received dental prophylaxis within 1 month prior to the Baseline visit;
* Oral pathology or a history of allergy to testing products;
* Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study; to be defined by the dental examiner;
* Subject participating in any other clinical study;
* Subject pregnant or breastfeeding;
* Subject allergic to oral care products, personal care consumer products, or their ingredients;
* Extended use of antibiotics or therapeutic mouthwash (eg: Chlorhexidine) any time during the three months prior to entry into the study;
* Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine);
* Current smokers and subjects with a history of alcohol or drug abuse;
* Subjects with orthodontic appliances or presence of fixed or removable prosthodontics dentures that may interfere with the evaluations
* An existing medical condition (eg: diabetic people) which prohibits eating or drinking for periods up to 4 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Löe-Silness Gingival Index | 21 days
  A Löe-Silness Gingival Index score from 0 to 3 will be assigned by the examining dentist to all scorable surfaces of the maxillary and mandibular teeth using a dental light and dental mirror. A whole mouth mean score for each subject will be determined by adding the values given by the examining dentist to each scorable surface and dividing that number by the total number of surfaces scored.

SECONDARY OUTCOMES:
Modified Quigley-Hein Plaque Index | 21 days
  The Turesky modification of the Quigley-Hein Plaque Index is a method for assessing dental plaque accumulation by scoring plaque presence on six surfaces of each tooth on a scale from 0 to 5.
Lobene Stain index | 21 days
  The labial/lingual surface of each tooth will be divided into two regions: the gingival region, and the body region. The gingival and body regions would be scored separately for yellow stains by use criteria for intensity or severity: 0- no stain, 1- light stain, 2-moderate stain, and 3-heavy stain. The extent to which these yellow stains covered the gingival and body regions will be scored: 0-no stain detected, only tooth color, 1- stain covering up to 1/3 of the region, 2- stain covering from 1/3 to 2/3 of the region, and 3- stain over two thirds of the region. The sum of the stain scores for a subject will be used as that subject's stain score.

CONTACTS AND LOCATIONS:
Overall Officials: Cassiano K Rosing, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No